CLINICAL TRIAL: NCT02527603
Title: Randomized Clinical Trial Comparing the Spaso Maneuver Versus the Self-assisted Boss-Holzach-Matter for Anterior Shoulder Dislocations
Brief Title: Spaso Versus Self-assisted Maneuver for Anterior Shoulder Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Francesc A. Marcano-Fernández, Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSPTCOT201501
Record Dates: First submitted 2015-08-15; First posted 2015-08-19 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Anti-Inflammatory Agents, Non-Steroidal; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spaso Method (Experimental): Randomized for Sp method + 1 initial dose of 50mg dexketoprofen IM or 25mg Oral
  Interventions: Procedure: Spaso method; Drug: Anti-Inflammatory Agents, Non-Steroidal
- Boss-Holzach-Matter Method (Experimental): Randomized for BHM method +1 initial dose of 50mg dexketoprofen IM or 25mg Oral
  Interventions: Procedure: Boss-Holzach-Matter method; Drug: Anti-Inflammatory Agents, Non-Steroidal

INTERVENTIONS:
Procedure: Boss-Holzach-Matter method — The patient holds both his hands around his knees in a supine position until the dislocated shoulder is reduced
  Other Names: Self-assited Method
  Arms: Boss-Holzach-Matter Method
Procedure: Spaso method — The physician holds the dislocated arm of the patient in a supine position and proceeds with gentle, soft movements of adduction, flexion and external rotation of the limb in this order until reduction is accomplished.
  Arms: Spaso Method
Drug: Anti-Inflammatory Agents, Non-Steroidal — All patients will be administered a dose of NSAI intra-muscular or orally ("Dexketoprofen", "Enantyum®") it is part of the normal treatment of these patients to cope with pain.
  Other Names: Pain Killer, "Enantyum®"

SUMMARY:
To compare the results and efficacy of the self-assisted Boss-Holzach-Matter maneuver for anterior shoulder dislocation and the Spaso method performed by a physician.

DETAILED DESCRIPTION:
Introduction: There are many described maneuvers in literature describing how to reduce an anterior shoulder dislocation. Most of these maneuvers are performed by a trained physician, however, seldom are these taught to patients in case of recurrence or accidental dislocations that may occur far from a trained professional to treat. The Boss-Holzach-Matter maneuver is a simple, easy to understand and easy to perform self assisted method that has not been compared to any other method.

Hypothesis: The Boss-Holzach-Matter method is a less painful maneuver compared to the Spaso method assuming an equal success rate.

Objective: To determine whether the Boss-Holzach-Matter method is a less painful method for anterior shoulder dislocations compares to the Spaso method assuming equal success rate.

Methodology: Fifty six patients presenting acute anterior shoulder dislocation will be randomized, at the time of the admission , to either Spaso reduction method performed by a physician or the self-assisted Boss-Holzach-Matter method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute anterior shoulder dislocation that are diagnosed in our hospital trauma area.

Exclusion Criteria:

* Fracture luxation of the same shoulder.
* Inability to cooperate due to mental or physical condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain that the patient experiences during the reduction procedure | Patients will be assessed throughout their visit to the Trauma Unit. No further following should be necessary.There will be no change in pain measurement, only the amount of pain felt during the manoeuvre.
  Pain the patient feels during the reduction maneuver. The patient will be asked after reduction to fill out a form with a analog visual scale with scores ranging from 0 [no pain] to 10 [worst possible pain].

CONTACTS AND LOCATIONS:
Overall Officials: David Marti, PhD, Study Director — Doctor
Locations (1):
- Corporación sanitaria Parc Taulí de Sabadell, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Sharing for other RCT, reviews, Meta analysis. Available from August 2017 Contact: famarcano@tauli.cat